CLINICAL TRIAL: NCT03398577
Title: Effects of SGLT2 Inhibitor on Markers of Inflammation, Atherosclerosis and Left Ventricular Strain in Diabetic Patients With Coronary Artery Disease
Brief Title: Effects of SGLT2 Inhibitor in Diabetic Patients With Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Robert Klempfner Heart Rehabilitation Institute, Proffesor Robert Kempfner, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SGLT2
Record Dates: First submitted 2017-12-21; First posted 2018-01-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Coronary Disease With Diabetes Mellitus
Keywords: Coronary disease; diabetes; SGLT2I; Inflammation Mediators
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: The study is designed as a single-center, double-blinded, placebo controlled, 2-arm clinical trial to provide evidence on the effects of Dapagliflozin on key biomarkers of athero-thrombosis, inflammation and ventricular loading conditions (NT ProBNP).
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Eligible patients (HbA1C ≥ 7% and ≤ 9%) , who were allocated to the Intervention group will receive Dapagliflozin 10 mg in addition to oral anti-diabetic medication administered prior to study enrollment.
  Interventions: Drug: Dapagliflozin 10 MG [Farxiga]
- Control group (Placebo Comparator): Eligible patients (HbA1C ≥ 7% and ≤ 9%) , who were allocated to the Control group will receive placebo in addition to oral anti-diabetic medication administered prior to study enrollment.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin 10 MG [Farxiga] — Computer based randomization software will be used in order to randomize eligible consenting subjects to placebo or Dapagliflozin 10 mg treatment using a 1:2 ratio.
  Other Names: Farxiga
  Arms: Intervention group
Drug: Placebo Oral Tablet — Computer based randomization software will be used in order to randomize eligible consenting subjects to placebo or Dapagliflozin 10 mg treatment using a 1:2 ratio.
  Arms: Control group

SUMMARY:
The aim of this study is to explore the effect of newly added SGLT2I medication or placebo, to standard medication regimen in diabetic patients with documented stable coronary disease. Therefore, in the present study the investigators plan to focus on possible anti-inflammatory and athero-thrombotic protective effects of Dapagliflozin compared to placebo, in secondary prevention population of stable coronary patients with diabetes. Additionally, the investigators will explore NT proBNP dynamics, which related to ventricular filling pressures in this specific population.

DETAILED DESCRIPTION:
Patients with ischemic heart disease and diabetes are at a particularly high risk for the recurrence of cardiovascular events, conversely, certain classes of oral anti-diabetic medications have been shown to cause hypoglycemia with adverse cardiovascular implications 1,2. Diabetes induces complex vascular changes, promoting accelerated atherosclerosis and a hyper-coagulable state, as can be assessed indirectly by a number of markers. Principal perturbations include endothelial dysfunction, increased inflammatory plaque infiltration, adhesion molecule over-expression and adverse effects of circulating fatty acids and advanced glycosylation end-products.

Cardiovascular safety of anti-diabetic medications is of paramount importance and has been under recent FDA and EDQM scrutiny. A number of hypoglycemic drugs, especially sulfonylureas, have been associated with significant hypoglycemia and adverse events induced by sympathetic activation. Activation of the sympathetic system has numerous implications, including surges of heart rate, blood pressure but also pro-inflammatory and pro-coagulant effects. This partially explains increased cardiovascular adverse events noted with these drugs. Newer classes of antidiabetic medication have recently shown improved survival outcomes in patients with cardiovascular disease, yet the exact mechanisms of the observed risk reduction are mostly yet to be elucidated 3,4. One possible mechanism is anti-inflammatory effect exerted directly or indirectly by SGLT2I or diuretic effect leading to left ventricular unloading with NT pro BNP level reduction.

The aim of this study is to explore the effect of newly added SGLT2I medication or placebo, to standard medication regimen in diabetic patients with documented stable coronary disease. Reduction of inflammatory marker levels is of great clinical importance and has been shown to correlate with reduction in significant clinical events5. Therefore, in the present study we plan to focus on possible anti-inflammatory and athero-thrombotic protective effects of Dapagliflozin compared to placebo, in secondary prevention population of stable coronary patients with diabetes. Additionally, the investigators will explore NT proBNP dynamics, which related to ventricular filling pressures in this specific population.

Key representative markers for the present study are chosen in order to correctly represent alterations in: inflammation (hs-CRP, IL(interleukin) -1 beta, IL-6, P-Selectin, TNF-alfa), and LV strain (NT pro BNP).

The effect of SGLT2I on the above-mentioned parameters has not been studied in humans. Accordingly, the demonstration of significant improvements in markers of athero-thrombosis and inflammation in high-risk diabetic patients is of great clinical importance and novelty that may be employed for the reduction of major cardiovascular events in this population.

Importantly, the effects of SGLT2I therapy will be evaluated in a prospective controlled clinical trial in a closely supervised cardiac rehabilitation setting, which includes lifestyle changes, regular, quantifiable physical activity, and predefined nutritional interventions.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus on oral therapy
* Stable documented ischemic Heart disease (> 60 days post AMI, CABG or PCI)
* Sub-optimal Hb A1c defined as ≥ 7%
* Age > 21
* Life expectancy >1 year

Exclusion Criteria:

* Events of clinical hypoglycemia during the past 6 months
* Recent (< 60 days) acute coronary syndrome (ACS) or Cerebrovascular accident
* Transient ischemic attack (TIA) within the past year.
* Significant renal impairment (eGFR < 60 ml/min/1.73 m2)
* History of recurrent UTI \ vaginitis
* Past bladder cancer (TCC or other)
* History of diabetic keto-acidosis
* Planned coronary intervention or planed surgical intervention (PCI or CABG)
* Unstable arrhythmias (i.e. rapid atrial fibrillation, symptomatic bradycardia, recurrent ventricular arrhythmia that are clinically significant, etc.)
* Known hypersensitivity to study drug
* Type I diabetes
* Current Hb A1c >9%
* Current Insulin treatment
* Active treatment with SGLT2I medication
* Inability to comply with study protocol
* Active malignancy other than basal cell carcinoma (BCC)
* Clinically advanced congestive heart failure - NYHA class III-IV
* Severe left ventricular dysfunction (LVEF<30%) with NYHA II or any NYHA class with documented recent heart failure decompensation (<3 months)
* Severe stable cardiac angina CCS III - IV or Unstable angina
* Chronic inflammation (i.e. IBD, Lupus, inflammatory arthritis, rheumatoid arthritis) or chronic infection (i.e. chronic diabetic foot infection)
* Pregnancy, lactation or child-bearing potential

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in interleukin (IL)-1β levels | 3 months
  Percent reduction in IL-1 β will be calculated as follows:(Baseline IL-1 minus follow-up [3-month] IL-1)/Baseline IL1; with value multiplied by 100.

SECONDARY OUTCOMES:
Percent reduction in additional biomarkers | 3 months
  Additional biomarkers including: IL-1 alpha, IL-8, IL-10, IL-17, tumor necrosis factor (TNF)-alpha, monocyte chemotactic protein (MCP-1) . Percent reduction will be calculated as mentioned above
Safety from events of clinical hypoglycemia | 3 Months
  Events of clinical hypoglycemia are defined as:
  palpitations, tremor, hunger, sweating and objective measurement of blood glucose ≤ 70 mg/dl
Reduction in BMI | 3 Months
  Changes in BMI will be calculated according to weight and height measurements at enrollment comparing to its value following 3-month active treatment period.
Reduction in HB A1c | 3 Months
  Reduction will be calculated by comparing HB A1c value at enrollment to its value following 3-month active treatment period.
NTpro BNP | 3 Months
  Changes in BNP will be calculated by comparing it's value at enrollment to its value following 3-month active treatment period.
MMP-9 percent reduction | 3 Months
  Percent reduction will be calculated as mentioned on outcome 1
Percent change in Adiponectin levels | 3 Months
  Percent reduction will be calculated as mentioned on outcome 1

CONTACTS AND LOCATIONS:
Overall Officials: Robert Klempfner, Proffesor, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Cardiac Rehabilitation Institute, Tel Litwinsky, Israel